CLINICAL TRIAL: NCT05153200
Title: Early Changes in Pain, Disease Activity, and Ultrasound Evidence of Inflammatory Synovitis in Patients Receiving JAK-inhibitor vs. TNF-inhibitor Therapy for Active Rheumatoid Arthritis: A Feasibility Study.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other); University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20210654-01H
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — upadacitinib; Adalimumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: MSK-US assessors will be blinded to treatment allocation, pain scores, and disease activity measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upadacitinib(Rinvoq) (Experimental): Upadacitinib(Rinvoq) 15 mg po daily
  Interventions: Drug: Upadacitinib
- Adalimumab(Idacio) (Active Comparator)
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Upadacitinib — 15 mg po daily
  Other Names: Rinvoq
  Arms: Upadacitinib(Rinvoq)
Drug: Adalimumab — 40 mg sc every other week
  Other Names: Idacio
  Arms: Adalimumab(Idacio)

SUMMARY:
The purpose of this phase 4 pilot study is to assess 1-year recruitment, and 6-month retention rates for participants with rheumatoid arthritis (RA) recruited to this study. Secondarily, we aim to study the difference in multifaceted pain scoring and Musculoskeletal Ultrasound (MSK-US)-detected synovitis between those treated with Upadacitinib vs Adalimumab.

DETAILED DESCRIPTION:
This is a 26-week phase 4 randomized, single-blind, parallel-group, active treatment-controlled pilot/feasibility study designed to primary assess recruitment and retention rates and to secondarily assess the efficacy of Upadacitinib vs Adalimumab in controlling multiple measures of pain and MSK-US-detected synovitis in those with Active Rheumatoid Arthritis.

Participants with active RA despite combination conventional synthetic Disease Modifying Antirheumatic Drugs (csDMARD), alternative biologic DMARD (bDMARD), or alternative targeted synthetic DMARD (tsDMARD) will be randomized in a 1:1 ratio to:

* Upadacitinib(Rinvoq) 15 mg orally (po) daily or
* Comparison Group: Adalimumab(Idacio) 40 mg subcutaneously (sc) every other week Baseline methotrexate may be continued if patient is receiving at time of study enrollment.

At 1 year after study initiation, recruitment rate over the first year will be measured and rate of 6-month participant retention will also be measured.

At baseline, 1 month, 3 months, and 6 months after initiation of study drug, disease activity, pain, MSK-US synovitis, and other patient important outcomes will be collected.

The study will be completed after 6-months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA based on ACR/EULAR 2020 Classification Criteria
* Moderate-to-high disease activity according to clinical disease activity indices
* Referred to the biologics clinic (The Ottawa Hospital Arthritis Centre) by their primary rheumatologist who practices within the division following decision to escalate to, or switch between, advanced therapy.

Exclusion Criteria:

* Any contraindication to initiation of either Upadacitinib or Adalimumab
* Unable to come to follow-up at 1, 3, and 6 months
* Current or planned (within 6 months) pregnancy or breastfeeding
* Inability to give informed consent
* Inability to communicate verbal or written responses to pain questionnaires
* Intraarticular steroid injections if done within 30 days of first visit
* Initiation of study intervention prior to baseline assessment
* Previous use of either study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 1 year
  Number of participants recruited to study
Retention Rate | 6 months
  Proportion of participants who complete the 6 months of follow-up

SECONDARY OUTCOMES:
Change in 100 mm Pain visual analogue scale (VAS) | 6 months
  "no pain" and "pain as bad as it can be" as anchors (MCID=11 mm)
Change in McGill Pain Questionnaire (MPQ) | 6 months
  Detailed assessment of pain quantity, quality, and impact (MCID=5)
Change in Widespread Pain Index (WPI) | 6 months
  Score of 4 or more indicates widespread pain (no known MCID)
Change in PainDETECT Questionnaire (PDQ) | 6 months
  Nociceptive (PDQ<13, unclear pain PDQ 14-18, neuropathic pain >18)
Change in OMERACT (Outcome Measures in Rheumatoid Arthritis in Clinical Trials) ultrasound task force Global Synovitis Score (GLOESS). | 6 months
  US assessment of 32 joints assessing for Gray-scale synovitis and power-Doppler findings.
Change in Swollen Joint Count (44) | 6 months
Change in Tender Joint Count (44) | 6 months
Change in Physician Global Assessment of Disease Severity | 6 months
  VAS
Change in Patient Global Assessment of Disease Severity | 6 months
  VAS
Change in Health Assessment Questionnaire | 6 months
American College of Rheumatology (ACR) 20 response | 6 months
ACR 50 response | 6 months
ACR 70 response | 6 months
Change in Erythrocyte Sedimentation Rate | 6 months
Change in C-Reactive Protein | 6 months
Change in Disease Activity Score (DAS)-28-ESR | 6 months
Change in DAS-28-CRP | 6 Months
Change in Clinical Disease Activity Index (CDAI) | 6 months
Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT) | 6 months
Change in Insomnia Severity Index (ISI) | 6 months
Change in Short Form 36 (SF-36) | 6 months
Change in Patient Health Questionnaire (PHQ-9) | 6 months
Adverse Events | 6 months
Serious Adverse Events | 6 months
Drop-out due to Adverse Events | 6 months

IPD SHARING:
Plan to Share IPD: No